## The Feasibility Study of The Delivery of The Book From Self Help Plus: "Doing What Matters in Times of Stress: An Illustrated Guide"

[NCT ID not yet assigned]

12/11/2020

## **Study Protocol**

A feasibility study will be conducted to see if it is realistic or feasible to test the effectiveness the Doing What Matters in Times of Stress: An Illustrated Guide for Turkish and Syrian individuals with psychological stress. Participants will be recruited through the advertisement of the study on social media. Potential participants who applies to participate in the study will complete an online screening & baseline survey if they approve the online informed consent form.

The screening questionnaire will include Kessler Psychological Distress Scale (K10) and a suicidality screening form. The baseline questionnaire will include Patient Health Questionnaire-9 (PHQ-9), General Anxiety Disorder-7 (GAD-7), four items from PTSD Checklist for DSM-5 (PCL-5), an item from the World Health Organization Quality of Life (WHOQOL), the General Self-Efficacy Scale and the Acceptance and Action Questionnaire (AAQ-2). The participants who are older than 18 years old, who are literate, scores 15 or above from K10 and who does not have imminent suicidal risk will be included in the study. At the end, we aim to include 128 (64 Turkish and 64 Syrian individuals) participants in the study. The participants will be randomized into intervention and control arm.

The participants' phone numbers and e-mail addresses will be received within the survey. The booklet will be sent to the participants in the intervention arm. The psychologists who are trained on delivering Doing What Matters in Times of Stress: An Illustrated Guide will get in contact with the participants three times during the participants. For the first time, psychologists will inform the participants about the program and introduce the booklet. For the second time, the psychologists will get in contact with the participants to see whether they need any support in using the booklet. And for the third and last time, psychologists will get in contact to review the process with the participants and get feedback. The booklet consists of five sections and related audio recordings. The participants will be asked to work on each section for a week. The whole program will take five weeks. The psychologists will call the participants during the first week, third week and the fifth week.

The participants will receive another online survey link one week after the completion of the program. The post test will include the same questionnaires with the pre-assessment. After the post-assessments are completed, the participants in the control group will also receive the booklet and the audio recordings.

Data will be analyzed by using a statistical package called IBM SPSS 21.0. Considering the groups as fixed factor, linear mixed models will be used to evaluate the effectiveness of SH+ intervention on primary (PHQ-9) and secondary outcomes (GAD-7, PCL-5, WHOQOL, General Self-Efficacy, AAQ-2).